CLINICAL TRIAL: NCT06694077
Title: Comparative Study of Dexamethasone Plus Bupivacaine Versus Bupivacaine in Suprazygomatic Maxillary Nerve Block for Management of Postoperative Pain in Adenotonsillectomy Patients
Brief Title: Suprazygomatic Maxillary Nerve Block for Management of Postoperative Pain in Adenotonsillectomy Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub saad kamal kamel, Resident at anaesthesia and icu, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-2024-200938
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Tonsillectomy Postoperative Adverse Events; Dexamethasone Administration; Bupivacaine
MeSH Terms: interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine with Dexamethasone (Experimental): bilateral suprazygomatic maxillary nerve block will be performed with 1 mL of 0.5% bupivacaine was added to 0.1 mg.kg-1 dexamethasone and diluted to 2 mL with 0.9% saline.
  Interventions: Drug: Bupivacaine with Dexamethasone
- Bupivacaine only (Experimental): bilateral suprazygomatic maxillary nerve block will be performed with 1 mL of 0.5% bupivacaine alone and diluted to 2 mL with 0.9% saline
  Interventions: Drug: Bupivacaine only

INTERVENTIONS:
Drug: Bupivacaine with Dexamethasone — bilateral suprazygomatic maxillary nerve block will be performed with 1 mL of 0.5% bupivacaine was added to 0.1 mg.kg-1 dexamethasone and diluted to 2 mL with 0.9% saline.
  Arms: Bupivacaine with Dexamethasone
Drug: Bupivacaine only — bilateral suprazygomatic maxillary nerve block will be performed with 1 mL of 0.5% bupivacaine alone and diluted to 2 mL with 0.9% saline
  Arms: Bupivacaine only

SUMMARY:
This study explores the effectiveness of adding dexamethasone to a suprazygomatic maxillary nerve block for postoperative pain relief in children undergoing adenotonsillectomy. The procedure, often performed to address recurrent infections and airway obstruction, results in significant pain due to inflammation and nerve irtypicallyritation. Traditional pain management methods, such as systemic analgesics, may be inadequate or lead to side effects in children. By combining dexamethasone, a potent anti-inflammatory, with local anesthetics, this trial aims to determine if enhanced pain control and a reduction in opioid use can be achieved.

The randomized, double-blind clinical trial will involve 80 children aged 3 to 10 years, randomized into two groups: one receiving the nerve block with bupivacaine and dexamethasone, and the other receiving bupivacaine alone. Pain will be assessed postoperatively using the FLACC score, with secondary measures including time to first analgesia, total analgesic use, hemodynamic stability, and any complications.

This study aims to demonstrate that the addition of dexamethasone may provide superior pain management in pediatric adenotonsillectomy, offering a safer, opioid-sparing alternative for postoperative care.

DETAILED DESCRIPTION:
This study is about the Analgesic Effect of Suprazygomatic Maxillary Nerve Block with and without Dexamethasone in Pediatric Adenotonsillectomy: A Randomized Double-Blinded Clinical Trial," investigates the effectiveness of adding dexamethasone to a suprazygomatic maxillary nerve block for postoperative pain management in children undergoing adenotonsillectomy. Adenotonsillectomy, a frequent surgical procedure in pediatric patients to address chronic infections and airway obstruction, is commonly associated with significant postoperative pain due to thermal and mechanical injury to tissues. This injury triggers inflammation, muscle spasms, and nerve irritation, which can lead to severe discomfort, decreased oral intake, and potential complications like dehydration.

The tonsils are primarily innervated by the maxillary division of the trigeminal nerve and the glossopharyngeal nerve, while the adenoids are innervated by branches of the trigeminal nerve alone. Despite traditional systemic analgesics being standard in pain management for such cases, they may not always provide adequate relief and can introduce undesirable side effects, particularly in pediatric patients. This limitation has spurred interest in regional anesthesia techniques, such as the suprazygomatic maxillary nerve block, which has been used in various facial and dental procedures but is less common in adenotonsillectomy. Combining dexamethasone, a potent corticosteroid known for its anti-inflammatory properties, with local anesthetics could provide enhanced analgesia and prolong the block's duration, potentially reducing the need for additional opioids post-surgery.

This randomized, double-blind, controlled clinical trial will be conducted at the ENT Operating Theatre at Assiut University Hospitals. The study will involve 80 pediatric patients between 3 and 10 years old, classified as ASA physical status I or II, who are scheduled for adenotonsillectomy. Participants will be randomized into two groups of 40 each: Group A will receive a suprazygomatic maxillary nerve block with 0.5% bupivacaine combined with dexamethasone, and Group B will receive the same nerve block with bupivacaine alone.

For statistical analysis, data will be verified, coded, and processed using IBM-SPSS 24.0 software. Mean and standard ddeviations will be calculated for normally distributed variables, and a two-way repeated measures ANOVA will be used to analyze pain score trends over time. A significance level of p<0.05 will be used for all analyses.

Ultimately, this study aims to establish whether adding dexamethasone to the suprazygomatic maxillary nerve block could enhance pain control, reduce the need for systemic analgesics, and improve overall recovery outcomes for pediatric patients undergoing adenotonsillectomy. Positive findings may position this combination as a safer, more effective pain management strategy, potentially improving the postoperative experience and outcomes in pediatric surgeries

ELIGIBILITY:
Inclusion Criteria:

* Parturient of American Society of Anesthesiologists (ASA) class I or II physical status
* Children scheduled for tonsillectomy with adenoidectomy

Exclusion Criteria:

* Patient's guardian refusal to participate in the study. Children with Behavioural changes; physical or developmental delay; neurological disorder or psychological disorder.
* Children on sedative or anticonvulsant medication.
* Bleeding diathesis
* History of sleep apnea
* Significant organ dysfunction, cardiac dysrhythmia, congenital heart disease
* Known allergy to the study drugs.
* Skin lesions or wounds at the puncture site of the proposed block

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
the total amount of analgesic requirements during first the 24hr after two different blocks. | Postoperative 24 hours

SECONDARY OUTCOMES:
Postoperative pain score, Faces, Legs, Activity, Cry, Consolability (FLACC) | 1hour , 2hour, 6hour, 12hour, 24hour

IPD SHARING:
Plan to Share IPD: No